CLINICAL TRIAL: NCT06757257
Title: Special Drug Use-results Survey for Long-term Use (Fostamatinib)
Status: Recruiting | Type: Observational
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TLPMS01
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fostamatinib treatmented
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — oral administration

SUMMARY:
The purpose of this survey is evaluating the safety and efficacy of long-term administration of fostamatinib for Japanese patients with chronic idiopathic thrombocytopenic purpura under actual conditions of use.

DETAILED DESCRIPTION:
The purpose of this survey is evaluating the safety and efficacy of long-term administration of fostamatinib for Japanese patients with chronic idiopathic thrombocytopenic purpura under actual conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic idiopathic thrombocytopenic purpura who are treatment with fostamatinib for the first time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic idiopathic thrombocytopenic purpura who are treatment with fostamatinib for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Tokyo and Japanese Other Cities, Japan

IPD SHARING:
Plan to Share IPD: No